CLINICAL TRIAL: NCT01125566
Title: LUX-Breast 1; An Open Label, Randomised Phase III Trial of BIBW 2992 and Vinorelbine Versus Trastuzumab and Vinorelbine in Patients With Metastatic HER2-overexpressing Breast Cancer Failing One Prior Trastuzumab Treatment
Brief Title: LUX-Breast 1: BIBW 2992 (Afatinib) in HER2-positive Metastatic Breast Cancer Patients After One Prior Herceptin Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.75; 2009-015476-98 (EudraCT Number)
Record Dates: First submitted 2010-05-10; First posted 2010-05-18 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Afatinib; Trastuzumab; Vinorelbine

ARMS (2):
- Arm B: trastuzumab with vinorelbine (Active Comparator): patients receive weekly intravenous infusion of trastuzumab and vinorelbine
  Interventions: Drug: trastuzumab; Drug: vinorelbine
- Arm A: BIBW 2992 with vinorelbine (Experimental): patients receive BIBW 2992 tablets once daily combined with weekly intravenous infusion of vinorelbine
  Interventions: Drug: BIBW 2992; Drug: vinorelbine

INTERVENTIONS:
Drug: BIBW 2992 — patients receive BIBW 2992 tablets once daily and can reduce dose for adverse event management
  Arms: Arm A: BIBW 2992 with vinorelbine
Drug: trastuzumab — patients receive trastuzumab 2mg/kg intravenously every week
  Arms: Arm B: trastuzumab with vinorelbine
Drug: vinorelbine — patients receive vinorelbine 25mg/m² intravenously every week
  Arms: Arm B: trastuzumab with vinorelbine
Drug: vinorelbine — patients receive vinorelbine 25mg/m² intravenously every week
  Arms: Arm A: BIBW 2992 with vinorelbine

SUMMARY:
To investigate the efficacy and safety of BIBW 2992 in combination with vinorelbine i.v. chemotherapy as treatment in patients with HER2-overexpressing, metastatic breast cancer, who failed one prior trastuzumab (Herceptin®) treatment

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed diagnosis of HER2-overexpression breast cancer
* Stage IV metastatic disease
* Must have progressed on one prior trastuzumab treatment
* no more than one prior trastuzumab based therapy regimen (either adjuvant or first-line)
* Must have received anthracycline and/or taxane based chemotherapy for adjuvant treatment of breast cancer or first-line treatment of metastatic breast cancer
* Must have (archived) tumour tissue sample available for central re-assessment of HER2-status
* At least one measurable lesion according to RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1 .

Exclusion criteria:

* Prior treatment with Epidermal Growth Factor Receptor/Human Epidermal Growth Factor Receptor(EGFR/HER2)-targeted small molecules or antibodies other than trastuzumab
* Prior treatment with vinorelbine
* Known pre-existing interstitial lung disease
* Active brain metastases
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to randomisation.
* Cardiac left ventricular function with resting ejection fraction of less than 50%.
* Patients unable to comply with the protocol.
* Any contraindications for therapy with vinorelbine or trastuzumab.
* Known hypersensitivity to BIBW 2992 or the excipients of any of the trial drugs.
* Use of any investigational drug within 4 weeks of randomisation.
* Inadequate hepatic, renal and haematologic organ function

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2010-06-22 (Actual); Primary Completion 2013-06-08 (Actual); Study Completion 2018-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (207):
- United States (14):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Robert A. Moss MD, FACP, Inc, Fountain Valley, California
  - St. Jude Heritage Healthcare, Fullerton, California
  - University of California, Los Angeles, California
  - Cancer Care Associates Medical Group, Inc, Redondo Beach, California
  - Santa Barbara Hematology Oncology Medical Group, Inc, Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - North Shore Cancer Research Associates, Skokie, Illinois
  - Cedar Valley Cancer Center, Waterloo, Iowa
  - Pro Health Care Associated, Lake Success, New York
  - Hope Women's Cancer Center, Asheville, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Utah Cancer Specialists Cancer Center, Salt Lake City, Utah
- Argentina (4):
  - Instituto Medico de Asistencia e Investigaciones S. A., Buenos Aires
  - Hospital Britanico, Capital Federal
  - Sanatorio de la Provodencia, Ciudad Autonoma de Bs As
  - Sanatorio Parque, Rosario
- Australia (5):
  - Port Macquarie Base Hospital (PMBH), Port Macquarie, New South Wales
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Peninsula Haematology & Oncology, Frankston, Victoria
  - Maroondah Hospital, Ringwood East, Victoria
  - Mount Medical Centre, Perth, Western Australia
- Austria (2):
  - Ordensklinikum Linz GmbH - Barmherzige Schwestern, Linz
  - Kaiser Franz Josef Spital Vienna, Vienna
- Belarus (4):
  - Grodno Regional Clinical Hospital, Grodno
  - Public Health Inst. Minsk City Clinical Oncology Dispensary, Minsk
  - N. N. Alexandrov National Cancer Center of Belarus, Minsk Region
  - Vitebsk Regional Clinical Oncology Dispensary, Vitebsk
- Belgium (3):
  - Brussels - HOSP Jules Bordet, Brussels
  - Edegem - UNIV UZ Antwerpen, Edegem
  - Liège - HOSP St-Joseph, Liège
- Brazil (9):
  - Centro de Pesquisas Clínicas em Oncología, Cachoeiro de Itapemirim
  - Hospital Santa Cruz, Curitiba
  - Associacao Hospital de Caridade de Ijui, Ijuí
  - Associação Hospitalar Moinhos de Vento, Porto Alegre
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Centro de Novos Tratamentos CliniOnco, Porto Alegre
  - Instituto Nacional do Câncer - INCA, Rio de Janeiro
  - Faculdade de Medicina do ABC, Santo André
  - Centro de Referência da Saude da Mulher-Hosp Perola Byington, São Paulo
- Canada (7):
  - BC Cancer Agency - Vancouver, Vancouver, British Columbia
  - Dr. Leon Richard Oncology Centre, Moncton, New Brunswick
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - CHU de Quebec-Universite Laval Research Centre, Québec
- Instituto Clínico Oncológico del Sur - ICOS, Temuco, Chile
- China (20):
  - Cancer Hospital of Chinese Academy of Medical Science, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - 307 Hospital of PLA, Beijing
  - Chinese PLA General Hospital, Beijing
  - First Hospital of Jilin University, Changchun
  - West China Hospital, Chengdu
  - Fujian Provincial Tumor Hospital, Fuzhou
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - NanFang Hosptial, Guangzhou
  - The Third Affiliated Hospital of Harbin Medical University, Haerbin
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Qilu Hospital, Shangdong University, Jinan
  - the 81th Hospital of PLA, Nanjing
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Wuhan Union Hospital, Wuhan
- Czechia (4):
  - Hospital Ceske Budejovice, České Budějovice
  - University Hospital Olomouc, Olomouc
  - General Faculty Hospital, Prague, Prague
  - MEDICON a.s., Praha 4, Prague
- Egypt (2):
  - Oncology Centre- Mansoura University, Al Mansurah
  - El Manial Specialized Hospital, Cairo
- France (12):
  - HOP Amiens-Picardie Sud, Amiens
  - CTR P Papin, Onco, Angers, Angers
  - HOP Jean Minjoz, Besançon
  - CLI Bordeaux Nord Aquitaine, Bordeaux
  - CTR J Perrin, Onco, Clermont-Ferrand, Clermont-Ferrand
  - HOP Victor Hugo, Le Mans
  - CTR Catherine de Sienne, Nantes
  - HOP Saint-Louis, Paris
  - INS Jean Godinot, Onco, Reims, Reims
  - CTR Eugène Marquis, Rennes
  - CTR René Huguenin, Saint-Cloud
  - CTR Paul Strauss, Strasbourg
- Germany (15):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Medizinisches Zentrum Bonn, Bonn
  - OnkoDok GbR, Bottrop
  - Universitätsklinikum Köln (AöR), Cologne
  - St. Elisabeth-Krankenhaus, Cologne
  - DONAUISAR Klinikum Deggendorf-Dingolfing-Landau gKU, Deggendorf
  - Universitätsklinikum Erlangen, Erlangen
  - Kliniken Essen - Mitte gGmbH, Essen
  - Gynäk.-onkol. Gem.praxis, Dr. Uleer, Hildesheim, Hildesheim
  - Universitätsklinikum Magdeburg AöR, Magdeburg
  - Klinikum der Universität München - Campus Innenstadt, München
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Onkologische Praxis Oldenburg, Oldenburg
  - Universitätsfrauenklinik am Klinikum Südstadt, Rostock
  - Facharzt für Innere Medizin, Wuppertal
- India (13):
  - Gujarat Cancer and Research Institute, Ahmedabad
  - Sujan Surgical Cancer Hospital, Amravati
  - KIDWAI memoraial Institute of oncology, Bangalore
  - Sri Venkateshwara Hospital, Bengaluru
  - Dr. Rai Memorial Cancer Centre, Chennai
  - Bibi General Hospital and Cancer Centre, Hyderabad
  - Orchid Nursing Home, Kolkata
  - Natinal Cancer Institute, Maharagama
  - Central India Cancer Research Institute, Nagpur
  - Curie Manavata Cancer centre, Nashik
  - Jehangir Hospital Oncology Department, Pune
  - K.E.M Hospital, Pune
  - King George Hospital, Visakhapatnam
- Ireland (4):
  - Beaumont Hospital, Dubliin 9
  - Mater Misericordiae University Hospital, Dublin
  - St James's Hospital, Dublin
  - St Vincent's University Hospital, Dublin
- Israel (5):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem 91031, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center Tel Hashomer, Tel Litwinsky
- Italy (3):
  - Azienda Ospedaliera Universitaria Arcispedale Sant'Anna, Ferrara
  - Istituto Europeo di Oncologia, Milan
  - P.O. Monserrato, Monserrato (CA)
- Japan (3):
  - Tokai University Hospital, Kanagawa, Isehara
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka, Osaka
  - National Cancer Center Hospital, Tokyo, Chuo-ku
- Latvia (2):
  - P. Stradins Clinical Univ. Hospital, Oncology Clinic, Riga
  - Riga East Univ. Hospital, Oncology Centre, Riga
- Hammoud Hospital University Medical Centre (HHUMC), Lebanon, Lebanon
- Lithuania (2):
  - Hospital of Lithuanian Univ.of HealthSciences Kauno Klinikos, Kaunas
  - National Cancer Institute, Vilnius, Vilnius
- Hospital de Jesus, Colonia Centro, Mexico
- Netherlands (6):
  - Albert SchweitzerZiekenhuis, Dordrecht
  - Máxima Medisch Centrum, locatie Eindhoven, Eindhoven
  - Zuyderland Medisch Centrum, Geleen
  - Zuyderland Medisch Centrum, Heerlen
  - METC Academisch Ziekenhuis Maastricht/Universiteit van Maastricht, Maastricht
  - Isala Zwolle, Zwolle
- Peru (4):
  - Hospital Nacional Adolfo Guevara Velasco, Cusco
  - Clinica San Judas Tadeo, Lima
  - Instituto Oncologico Miraflores S.A., Miraflores
  - Clinica Peruano Americana de Trujillo, Trujillo
- Poland (8):
  - Bialystock's Oncology Center, Bialystok
  - Wojewodzki Specialist Hospital No. 4, Bytom, Bytom
  - University Clinical Center, Gdansk, Gdansk
  - Provincial Specialist M. Kopernik Hospital, Lodz
  - Ziemia Lubelska Oncological Center, Lublin, Lublin
  - Oncology Centre of Olsztyn "KOPERNIK" Sp. z.o.o., Olsztyn
  - Wielkopolskie Oncology Centre n.a. Maria Sklodowska-Courie, Poznan
  - Military Medical Institute, Warsaw
- Portugal (5):
  - Instituto Português de Oncologia de Coimbra Francisco Gentil, Coimbra
  - CHUC, EPE - CHC-Maternidade Bissaya Barreto, Coimbra
  - IPO Lisboa Francisco Gentil, EPE, Lisbon
  - Centro Hospitalar São João,EPE, Porto
  - IPO Porto Francisco Gentil, EPE, Porto
- Russia (4):
  - St.Auton.Heal.Inst."Rep.Clin.Onc.Disp.of MoH of Rep. Tatarstan", Kazan'
  - N.A. Semashko Central Clinical Hospital, Moscow, Moscow
  - GUZ "Regional Clinical Oncology Dispensary", Ryazan
  - Regional Clinical Oncology Dispensary, Saint Petersburg
- Singapore (3):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
  - Johns Hopkins Singapore International Medical Center, Singapore
- Slovakia (3):
  - St. Jacobs Hosp.Outpat.Pneumology&Phthisiology Dept,Bardejov, Bardejov
  - National Institute of Oncology, Bratislava, Bratislava
  - POKO Policlinic Dept. of Clinical Oncology, Poprad
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- South Africa (6):
  - WCR CMJAH Clinical Trial Site, Johannesburg
  - Medical Oncology Centre of Rosebank, Johannesburg
  - GVI oncology Medi Clinic, Kraaifontein
  - Langenhoven Drive Oncology Centre, Port Elizabeth
  - Wilgers oncology, Pretoria
  - Rondebosch Oncology Centre, Rondebosch, Cape Town
- South Korea (6):
  - National Cancer Center, Goyang
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (8):
  - Hospital del Mar, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Complejo Hospitalario Universitario Insular - Materno Infantil, Las Palmas de Gran Canaria
  - Hospital Clínico San Carlos, Madrid
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Virgen de la Salud, Toledo
  - Hospital Arnau de Vilanova, Valencia
- Shatabdi Superspeciality Hospital, Maharashtra, Sri Lanka
- Taiwan (10):
  - Chang-Hua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipe Veterans General Hospital, Taipei
  - Koo Foundation Sun Yet-Sen Cancer Center, Taipei
  - Chang Gung Memorial Hospital(TaoYuan), Taoyuan
- Turkey (Türkiye) (2):
  - Hacettepe Universitesi Tip Fakultesi, Ic Hastaliklari ABD, Ankara
  - Ege Universitesi Tip Fakultesi Tibbi Onkoloji Bilim Dali, Izmir
- United Kingdom (4):
  - Ninewells Hospital & Medical School, Dundee
  - Guy's Hospital, London
  - The Royal Marsden Hospital, Sutton
  - Queen Elizabeth Hospital, Woolwich, London

REFERENCES:
- [Derived] Harbeck N, Huang CS, Hurvitz S, Yeh DC, Shao Z, Im SA, Jung KH, Shen K, Ro J, Jassem J, Zhang Q, Im YH, Wojtukiewicz M, Sun Q, Chen SC, Goeldner RG, Uttenreuther-Fischer M, Xu B, Piccart-Gebhart M; LUX-Breast 1 study group. Afatinib plus vinorelbine versus trastuzumab plus vinorelbine in patients with HER2-overexpressing metastatic breast cancer who had progressed on one previous trastuzumab treatment (LUX-Breast 1): an open-label, randomised, phase 3 trial. Lancet Oncol. 2016 Mar;17(3):357-366. doi: 10.1016/S1470-2045(15)00540-9. Epub 2016 Jan 26. PMID 26822398

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was randomised, active-controlled, open-label, parallel-group, 2 arm (2:1 ratio) trial in participants with metastatic human epidermal growth factor receptor 2 (HER2)-overexpressing breast cancer failing one prior trastuzumab treatment.
Pre-assignment Details: Participants were treated in the study until disease progression, undue toxicity, or withdrawal of consent. The cut-off date for RECIST-based efficacy was 08 Jun 2013; a second analysis (primarily for assessing Overall Survival (OS)) contains all data until final database lock (30 Jul 2018).
Groups:
- Afatinib + Vinorelbine (AV): Participants received oral treatment of film-coated Afatinib tablet at a starting dose of 40 milligram (mg) once daily and weekly 10 minutes intravenous infusion of Vinorelbine 25 mg/meter^2 (meter=m) on days 1, 8, 15, and 22 of each course. The treatment was administered in treatment courses of 28 days. For Afatinib, a protocol-defined dose-reduction scheme was to be followed if a participant experienced certain pre-specified adverse events. From 26 April 2013, any participant who had been randomised to the AV arm stopped treatment, had the option to switch to Trastuzamb + Vinorelbine.
- Trastuzumab + Vinorelbine (TV): Participants received an intravenous infusion of Trastuzumab 2 mg/kilogram (kg) weekly, following an initial loading dose of 4 mg/kg and weekly 10 minutes intravenous infusion of Vinorelbine 25 mg/m^2 on days 1, 8, 15, and 22 of each course. The treatment was administered in treatment courses of 28 days.
- AV Switched to TV: This group describes participants who discontinued AV treatment and switched to TV, provided they were without disease progression on AV, following data monitoring committee (DMC) recommendation to terminate recruitment on 26 April 2013.
Period: Patients Before the Switch (26Apr2013)
Arm/Group | Afatinib + Vinorelbine (AV) | Trastuzumab + Vinorelbine (TV) | AV Switched to TV
Started (Randomised) | 339 | 169 | 0
Treated | 337 | 169 | 0
Completed | 74 | 0 | 0
Not Completed | 265 | 169 | 0
Not completed — Progressive disease according to RECIST | 182 | 119 | 0
Not completed — Worsening of underlying cancer disease | 6 | 6 | 0
Not completed — Adverse Event | 25 | 5 | 0
Not completed — Protocol Violation | 0 | 2 | 0
Not completed — Refused to continue taking medication | 24 | 23 | 0
Not completed — Not treated | 2 | 0 | 0
Not completed — Other than listed above | 25 | 13 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Period: Patients Who Switched From AV to TV
Arm/Group | Afatinib + Vinorelbine (AV) | Trastuzumab + Vinorelbine (TV) | AV Switched to TV
Started | 0 | 0 | 75
Completed | 0 | 0 | 2
Not Completed | 0 | 0 | 73
Not completed — Progressive disease according to RECIST | 0 | 0 | 59
Not completed — Refused to continue taking medication | 0 | 0 | 7
Not completed — Worsening of underlying cancer disease | 0 | 0 | 3
Not completed — Other than listed above | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The TS included all randomised participantsbwho were documented to have taken at least 1 dose of study medication (i.e. afatinib, trastuzumab, or vinorelbine). One centre with 6 subjects was excluded from analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib + Vinorelbine (AV) | Trastuzumab + Vinorelbine (TV) | Total
Number analyzed (Participants) | 332 | 168 | 500
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.8 (11.3) | 53.1 (12.3) | 52.2 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 332 | 168 | 500
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data was not reported for this trial.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 172 | 81 | 253
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 136 | 72 | 208
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as time from randomisation to disease progression or death whichever occurs first. Assessed by investigator according to the Response Evaluation Criteria in Solid Tumours (RECIST 1.1). RECIST is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize") or worsen ("progress") during treatment.
  Only data collected until the cut-off date for RECIST 1.1 based endpoints (08Jun2013) were considered.
  Progression of disease was determined if at least 1 of the following criteria applied:
  * At least a 20% increase in the sum of the diameters (SoD) of target lesions taking as reference the smallest SoD recorded since the treatment started, together with an absolute increase in the SoD of at least 5 mm
  * Appearance of 1 or more new lesions
  * Unequivocal progression of existing non-target lesions
Time Frame: From randomization (07Sep2010) until disease progression, death or data cut-off (08Jun2013); Up to 34 months
Population: Randomised set (RS): The randomised set included all participants who were randomised to receive treatment, whether treated or not.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Afatinib + Vinorelbine (AV) | Trastuzumab + Vinorelbine (TV)
Number analyzed (Participants) | 339 | 169
Months | 5.49 [3.55 to 9.07] | 5.55 [3.55 to 10.84]
Statistical Analysis 1: Comparison: Afatinib + Vinorelbine (AV) vs Trastuzumab + Vinorelbine (TV); Test type: Superiority or Other; p = 0.4224, Regression, Cox — Two sided p-value was derived from a log rank test stratified by the setting of prior Trastuzumab failure, hormone receptors status and region of the investigational site; Hazard Ratio (HR) = 1.10, 95% CI [0.87 to 1.41] — Hazard ratio is derived from Cox proportional hazard model stratified by prior Trastuzumab failure, hormone receptors status and region of the investigational site

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from randomisation to death irrespective of the cause of the death.
  For patients who had not died up to the cut-off date (03Sep2013), the date they were last known to be alive was derived from the patient status records, the trial completion record, radiological imaging assessments, the study treatment termination record, and the randomisation date.
Time Frame: From randomisation (07Sep2010) to database lock (30Jul2018), up to 95 months.
Population: RS including participants with available data for OS.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Afatinib + Vinorelbine (AV) | Trastuzumab + Vinorelbine (TV)
Number analyzed (Participants) | 339 | 169
Months | 20.17 [10.74 to 39.52] | 29.60 [13.34 to 43.99]
Statistical Analysis 1: Comparison: Afatinib + Vinorelbine (AV) vs Trastuzumab + Vinorelbine (TV); Results of presented analyses are to be seen as exploratory (no confirmatory testing was performed); Test type: Superiority or Other; p = 0.0240, Regression, Cox — Two sided p-value from a log rank test stratified by the setting of prior Trastuzumab failure, hormone receptors status and region of the investigational site; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [1.03 to 1.63] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Best RECIST Assessment
Description: Best RECIST assessment is defined as CR, PR, stable disease (SD), progressive disease (PD) or not evaluable by investigator (RECIST version 1.1).
  CR for target lesions (TL): Disappearance of all target lesions.
  CR for non-target lesions (NTL): Disappearance of all non-target lesions and normalization of tumour marker level. All lymph nodes must be non-pathological in size (<10mm short axis).
  PR: At least a 30% decrease in the sum of diameters (SoD) of target lesions taking as reference the baseline sum diameters.
  SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as references the smallest SoD while on study.
  PD: At least a 20% increase in the SoD of target lesions, taking as references the smallest sum on study (this includes the baseline sum if that is the smallest on study). Also, the sum must also demonstrate an absolute increase of a least 5mm. Appearance of one or more new lesions.
Time Frame: From randomization (07Sep2010) until disease progression, death or data cut-off (08Jun2013); Up to 34 months
Population: RS including participants with available data for best RECIST assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib + Vinorelbine (AV) | Trastuzumab + Vinorelbine (TV)
Number analyzed (Participants) | 334 | 168
Percentage of participants
  Complete response (CR) | 3.3 | 3.0
  Partial response (PR) | 43.1 | 44.0
  Stable disease (SD) | 31.7 | 26.8
  Progressive Disease (PD) | 12.6 | 17.9
  Missing | 9.3 | 8.3
Statistical Analysis 1: Comparison: Afatinib + Vinorelbine (AV) vs Trastuzumab + Vinorelbine (TV); Results of presented analyses are to be seen as exploratory (no confirmatory testing was performed); Test type: Superiority or Other; p = 0.6431, Regression, Logistic; Logistic regression stratified by prior Trastuzumab failure, hormone receptors status and region of the investigational site; Odds Ratio (OR) = 1.090, 95% CI [0.756 to 1.572] — The odds ratio for the comparison afatinib + vinorelbine vs. trastuzumab + vinorelbine below 1 favours Afatinib

4. Secondary Outcome: Objective Response (OR)
Description: OR is defined as complete response (CR) and partial response (PR). Assessed by investigator according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1. Complete Response (CR) for target lesions (TL): Disappearance of all target lesions.
  Complete Response (CR) for non-target lesions (NTL): Disappearance of all non-target lesions and normalization of tumour marker level. All lymph nodes must be non-pathological in size (<10mm short axis)
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters.
  Other factors which add to the overall response of an imaging timepoint as PR are as below:-
  * CR in TL, but non-CR/Non-PD in NTL leads to PR
  * CR in TL, but not evaluated NTL leads to PR
  * PR in TL, but non-PD NTL or not all evaluated NTL leads to PR
Time Frame: Post baseline tumour-imaging was performed at Week 8, 16, 24, 32, 40, 48, 56 and then every 12 weeks (Until final data-base lock on 30 Jul 2018; Up to 95 months)
Population: RS including participants with available data for OR.
Measure: Number; unit: Percentage of participants (%)
Arm/Group | Afatinib + Vinorelbine (AV) | Trastuzumab + Vinorelbine (TV)
Number analyzed (Participants) | 334 | 168
Percentage of participants (%) | 46.4 [0.410 to 0.519] | 47.0 [0.393 to 0.549]
Statistical Analysis 1: Comparison: Afatinib + Vinorelbine (AV) vs Trastuzumab + Vinorelbine (TV); Results of presented analyses are to be seen as exploratory (no confirmatory testing was performed); Test type: Superiority or Other; p = 0.8829, Regression, Logistic; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.029, 95% CI [0.707 to 1.496] — The odds ratio for the comparison afatinib + vinorelbine vs. trastuzumab + vinorelbine below 1 favours AV

ADVERSE EVENTS:
Time Frame: From first administration of treatment within the trial until last administration of treatment within the trial, up to 76 months.
Description: Treated set was used for reporting the other adverse event and serious adverse event.
Arm/Group | Afatinib + Vinorelbine (AV) | Trastuzumab + Vinorelbine (TV) | AV Switched to TV
All-Cause Mortality (participants affected / at risk) | 235/337 | 111/169 | 3/75
Serious Adverse Events (participants affected / at risk) | 123/337 | 45/169 | 15/75
Other Adverse Events (participants affected / at risk) | 331/337 | 163/169 | 64/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib + Vinorelbine (AV) (N=337) | Trastuzumab + Vinorelbine (TV) (N=169) | AV Switched to TV (N=75)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 21 | 7 | 2
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 18 | 4 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 1
Keratitis (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 21 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhagic ascites (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 10 | 3 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 2 | 1 | 0
Catheter site inflammation (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Condition aggravated (General disorders) | 0 | 1 | 0
Device related thrombosis (General disorders) | 1 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 2 | 1 | 0
Mucosal inflammation (General disorders) | 5 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 15 | 5 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Abscess intestinal (Infections and infestations) | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0
Cardiac infection (Infections and infestations) | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 4 | 2 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Genital infection (Infections and infestations) | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 2 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Lymphangitis (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 2
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 4 | 2 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 1 | 0
Viraemia (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 3 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 5 | 3
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 2 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0
Gliosis (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Breast operation (Surgical and medical procedures) | 1 | 0 | 0
Central venous catheterisation (Surgical and medical procedures) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Shock (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib + Vinorelbine (AV) (N=337) | Trastuzumab + Vinorelbine (TV) (N=169) | AV Switched to TV (N=75)
Anaemia (Blood and lymphatic system disorders) | 103 | 62 | 25
Bone marrow failure (Blood and lymphatic system disorders) | 18 | 11 | 5
Leukopenia (Blood and lymphatic system disorders) | 115 | 68 | 28
Neutropenia (Blood and lymphatic system disorders) | 256 | 139 | 46
Abdominal pain (Gastrointestinal disorders) | 40 | 16 | 1
Abdominal pain upper (Gastrointestinal disorders) | 34 | 14 | 5
Constipation (Gastrointestinal disorders) | 35 | 27 | 6
Diarrhoea (Gastrointestinal disorders) | 270 | 45 | 7
Dyspepsia (Gastrointestinal disorders) | 16 | 12 | 3
Mouth ulceration (Gastrointestinal disorders) | 40 | 5 | 1
Nausea (Gastrointestinal disorders) | 102 | 47 | 6
Stomatitis (Gastrointestinal disorders) | 87 | 19 | 4
Vomiting (Gastrointestinal disorders) | 85 | 22 | 5
Asthenia (General disorders) | 63 | 25 | 5
Chills (General disorders) | 10 | 9 | 3
Fatigue (General disorders) | 106 | 51 | 10
Mucosal inflammation (General disorders) | 82 | 15 | 4
Oedema peripheral (General disorders) | 11 | 11 | 1
Pain (General disorders) | 23 | 7 | 2
Pyrexia (General disorders) | 74 | 32 | 11
Conjunctivitis (Infections and infestations) | 12 | 4 | 4
Influenza (Infections and infestations) | 7 | 0 | 4
Nasopharyngitis (Infections and infestations) | 30 | 11 | 2
Paronychia (Infections and infestations) | 63 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 32 | 27 | 8
Urinary tract infection (Infections and infestations) | 35 | 15 | 4
Alanine aminotransferase increased (Investigations) | 24 | 16 | 7
Aspartate aminotransferase increased (Investigations) | 22 | 11 | 8
Haemoglobin decreased (Investigations) | 28 | 6 | 5
Neutrophil count decreased (Investigations) | 16 | 13 | 6
Weight decreased (Investigations) | 48 | 10 | 6
White blood cell count decreased (Investigations) | 23 | 3 | 5
Decreased appetite (Metabolism and nutrition disorders) | 98 | 31 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 43 | 7 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 8 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 15 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 11 | 10 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 27 | 16 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 12 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 34 | 18 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 20 | 3
Dizziness (Nervous system disorders) | 34 | 18 | 5
Headache (Nervous system disorders) | 47 | 25 | 10
Hypoaesthesia (Nervous system disorders) | 9 | 11 | 2
Neuropathy peripheral (Nervous system disorders) | 15 | 16 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 15 | 11 | 2
Insomnia (Psychiatric disorders) | 26 | 28 | 3
Dysuria (Renal and urinary disorders) | 21 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 27 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 | 15 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 58 | 6 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 30 | 9 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 20 | 10 | 5
Acne (Skin and subcutaneous tissue disorders) | 22 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 34 | 13 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 45 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 20 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 42 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 31 | 8 | 2
Rash (Skin and subcutaneous tissue disorders) | 160 | 19 | 8

LIMITATIONS AND CAVEATS:
The Data Monitoring Committee recommended termination of recruitment due to low likelihood of the study meeting its primary objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.>